CLINICAL TRIAL: NCT02640846
Title: Potential Differences Between Levosimendan and Milrinone on Myocardial and Hemodynamic Variables in Patients With Septic Cardiomyopathy. Effects of Norepinephrine on Right Ventricular Function in Patient With Septic Shock.
Brief Title: Effects of Levosimendan, Milrinone and Norepinephrine on Left and Right Ventricular Function in Septic Shock
Acronym: SCLM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Keti Dalla, MD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: K050711
Record Dates: First submitted 2015-12-06; First posted 2015-12-29 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2015-12

CONDITIONS: Septic Shock; Cardiomyopathy
Keywords: Levosimendan; Milrinone; Myocardial strain; Septic cardiomyopathy; Norepinephrine
MeSH Terms: conditions — Shock, Septic; Cardiomyopathies | interventions — Norepinephrine; Milrinone; Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Norepinephrine (Active Comparator): Doser
  Interventions: Drug: Norepinephrine
- Milrinone (Active Comparator): Doser
  Interventions: Drug: Milrinone
- Levosimendan (Active Comparator): Doser
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Norepinephrine — Norepinephrine will be given to the patient due to septic shock. After the inclusion we will change the dose of Norepinephrine to achieve 3 different MAP-levels, 60 mmHg, 75 mmHg and 90 mmHg.
  Arms: Norepinephrine
Drug: Milrinone — Corotrope will be given and after 30 minutes of treatment the cardiac function will be assessed with echocardiography and systemic hemodynamics.
  Other Names: Corotrope
  Arms: Milrinone
Drug: Levosimendan — Levosimendan will be given and after 30 minutes of treatment the cardiac function will be assessed with echocardiography and systemic hemodynamics.
  Other Names: Simdax
  Arms: Levosimendan

SUMMARY:
The aim of this study is to investigate the effects milrinon and levosimandan on n heart function in septic cardiomyopathy and how norepinephrine affects the left and right ventricular function in patients with septick shock using pulmonary artery catheter, conventional and strain echocardiography.

DETAILED DESCRIPTION:
This is a prospective study where 30 patients with septic chock during the care in ICU, will be included. Patients with a history of previous heart disease are excluded from the study. Each patient is in need of norepinephrine infusion and on mechanical ventilation. Initially the mean arterial pressure (MAP) is randomly changed from 60 to 75 and then to 90 mmHg. Hemodynamic variables as blood pressure, cardiac output, pulmonary artery occlusion pressure (PAOP) will be registerd at each MAP-level, arterial line and pulmonary artery catheter (PAC) and the cardiac function will be assessed with conventional and strain echocardiography. Then, if the echocardiogram shows impaired LV-function will the patient be randomized to receive either Milrinone or Levosimendan. Hemodynamic variables as blood pressure, cardiac output, pulmonary artery occlusion pressure (PAOP) will be registered again, as well the cardiac function with conventional and strain echocardiography. Echocardiograms will be analysed for the determination of LV an RV strain. Potential differences between different levels of blood pressure as well as effects of Milrinone or Levosimendan on hemodynamic and echocardiographyc variables will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock.
* All patients will be resuscitated with fluids before the inclusion.
* Need of Norepinephrine infusion.
* Myocardial dysfunction in echocardiogram, either LVEF < 50% or Global Left Ventricular Systolic strain over -15%.

Exclusion Criteria:

* History of previous heart disease or pulmonary hypertension.
* Age < 18 years.
* Cardiac arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Changes in LV systolic strain | 1.5 hours
  Changes in LV systolic function (global strain) will be assessed by 2D speckle tracking echocardiography
Changes in RV systolic strain | 1.5 hours
  Changes in RV systolic function (RV free wall strain) will be assessed by 2D speckle tracking echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Erik Ricksten, Professor, Study Chair — Sahlgrenska Academy, dep of clinical science
Locations (1):
- Central intensivvårdsavdelning Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No